CLINICAL TRIAL: NCT03922646
Title: Neurocognitive Empowerment for Addiction Treatment (NEAT) in People With Opioid Use Disorder and Amphetamine Use Disorder: A Randomized Clinical Trial
Brief Title: Neurocognitive Empowerment for Addiction Treatment (NEAT) in Opioid Use Disorder and Amphetamine Use Disorder
Acronym: NEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-007
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Opioid-use Disorder; Amphetamine Use Disorders
Keywords: Cognitive Rehabilitation; Brain Rehabilitation; Treatment; Addiction; Heroin; Opiates; Meth; Methamphetamine
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEAT Active Experimental Group (Experimental): People in the active group will receive NEAT intervention
  Interventions: Behavioral: Neurocognitive Empowerment for Addiction Treatment (NEAT)
- Control Group (Active Comparator): People in the control group will receive non-essential regularly-scheduled programming (active control) coinciding with the same timeframe
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Neurocognitive Empowerment for Addiction Treatment (NEAT) — NEAT will be conducted in person, in groups of 6-14, and consist of 14, 1.5-hour sessions. Each NEAT session will consist of (1) a didactic, psychoeducation portion describing the concepts and skills of focus, (2) written material with descriptions of the concepts/skills in verbal and pictorial (cartoon) formats, (3) practicing with cognitive tasks relevant for each skill, (4) discussion of how they can monitor and practice each skill in their daily life. Specifically, we will provide psychoeducation, cognitive exercises, time-management and daily practice focused on domains of attention (focused and divided attention; attentional biases), memory (declarative, prospective, emotional memory), flexibility and inhibition, and problem-solving. Each session will discuss the relevance of these functions for the recovery from drug addiction and for managing affective/motivational symptoms commonly related to substance use (i.e., craving, anxiety, depression, trauma).
  Arms: NEAT Active Experimental Group
Behavioral: Active Control — The active control intervention will be composed of active, but non-essential aspects of the larger treatment program (i.e., those that treatment programs do not believe are necessary or central to their program, for example, art classes, exercise classes, chore time, or extra 12 steps meetings). This will ensure that subjects are not being prevented from accessing treatment that is already known to be helpful in substance use recovery, that the active control condition and NEAT intervention have equivalent credibility and expectancies, and optimizing the generalizability of findings.
  Arms: Control Group

SUMMARY:
Chronic drug addiction is not only associated with increased mental health symptoms, such as anxiety and depression, but also with brain (neural and cognitive) deficits. These neurocognitive deficits (NCDs) in memory, attention, decision-making, self-control and judgement disturb normal daily functioning and attempts for abstinence. These NCDs are also associated with worse long-term treatment outcomes. Current treatment programs for addiction to opioids and amphetamines are mainly focused on abstinence from illicit drugs with or without assistance of medications, with the assumption that these NCDs will subsequently heal. However, NCDs are found to persist even after a long-term abstinence and are thought to contribute to relapse, decreases quality of life, or lack of reintegration into society. Furthermore, NCDs (particularly related to attention and memory) are considered a potential obstacle for engagement in therapy services for addiction and associated mood, anxiety and trauma-related comorbidities (i.e., cognitive-behavioral therapies). Brain rehabilitation programs focused on compensatory strategies and training exercises for NCDs associated with traumatic brain injuries, stroke, multiple sclerosis and schizophrenia has consistently been found to improve functioning and long-term outcomes for these populations. There have been a few preliminary attempts to transplant cognitive rehabilitation with substance use populations, with some limited promise. However, these previous studies failed to link cognitive strategies with the drug use and affective/craving symptoms experienced by patients and also did not fully incorporate knowledge gained from neuroscientific research on opioid and/or methamphetamine addiction specifically.

The aim of this study is to characterize clinical efficacy for an intervention targeting NCDs in opioid and/or methamphetamine addiction by enhancing awareness and use of neurocognitive skills in the context of substance use recovery. This aim will be accomplished by randomizing 80 subjects with opioid and/or methamphetamine use disorder who are already enrolled in substance use treatment in the state of Oklahoma to also complete a novel "Neurocognitive Empowerment for Addiction Treatment" (NEAT) program developed by a group of investigators at Laureate Institute for Brain Research, Tulsa, Oklahoma. NEAT will be novel in (a) its use of cartoons, brain awareness games and real-life scenarios to ensure it is interactive and engaging, (b) the focus on the role of neurocognitive deficits in recovery from substance use and co-occurring mental health symptomatology, and (c) its incorporation of neuroscientific findings specific to substance use to the training and exercise strategies. Subjects will be followed up for twelve months after starting the program with different measures for addiction and mental health recovery to explore the efficacy of NEAT compared to the control intervention. Using LIBR's cutting-edge neuroimaging facilities before and after interventions, this study has the unique opportunity to monitor not only clinical outcomes but also potential changes NEAT may have on brain structure and function. In case of finding reasonable clinical efficacy for NEAT, it will be hopefully integrated as a manualized brain rehabilitation program to the substance use treatment programs.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in an established substance use treatment program, such as the Women in Recovery or 12&12 programs, Oxford Houses or others to be identified in the region) and diagnosed with Opioid Use Disorder and/or Amphetamine Use Disorder based on DSM V criteria using MINI structured interview.
2. Able to provide written informed consent.
3. Have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.
4. Completion of at least an 8th grade education, to help facilitate ability to engage in the written materials included in the NEAT program.
5. Current mental or physical health symptoms that require immediate attention (such as suicidal ideation with intent or plan; active psychotic symptoms; delirium; etc.)

Exclusion Criteria:

1. Unwillingness or inability to complete any of the major aspects of the study protocol, including self-report or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task).
2. Non-correctable vision or hearing problems.

For individuals to complete the brain imaging portion of the project, the following additional exclusion criteria will be used:

1. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
2. Current use of a medication or change in the dose or prescription of a medication within the 6 weeks prior to enrolling in the study that could potentially affect brain functioning (e.g., stimulants, antidepressants, anxiolytics, antipsychotics, mood stabilizers, anti-hypertensives). Inclusion of individuals reporting other types of medications or supplements not listed or considered thus far will be at the discretion of the PI according to evidence in the literature of it affecting brain function or brain blood flow.
3. Taking drugs that affect the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, excessive caffeine intake > 1000 mg/day).
4. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.
5. Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Change in craving self-report measured with Obsessive Compulsive Drug Use Scale (OCDUS) total score | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)

SECONDARY OUTCOMES:
Change in cognitive concerns self-report as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Concerns | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)

OTHER OUTCOMES:
Change in momentary drug craving self-report as measured with DDQ from before to after Intervention | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
  Desire for Drug Questionnaire (DDQ) has two subscores "desire and intention" (DI) and "negative reinforcement" (NR) subscores of the (Franken, et al., 2002).
Change in depression as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Depression | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in anger as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Anger | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in impulsive behavior as measured by UPPS Impulsive Behavior Scale | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
  UPPS (Urgency, Remediation, Perseverance, and Sensation Seeking) assesses an additional personality pathway to impulsive behavior, Positive Urgency, in addition to the four pathways assessed in the original version of the scale-- Urgency (now Negative Urgency), (lack of) Premeditation, (lack of) Perseverance, and Sensation Seeking.
Change in emotion regulation as measured by Difficulties in Regulation Scale (DERS) | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in positive affect as measured by NIH Toolbox Positive Affect | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in motivation as measured by NIH Toolbox Meaning and Purpose Survey | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in self efficacy in copying with stress as measured by NIH Toolbox Self-Efficacy (stress) | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in self efficacy in copying with chronic disease as measured by NIH Toolbox Self-Efficacy (chronic disease) | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in disability as measured by WHO Disability Assessment Schedule (WHODAS) | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in work and health performance as measured by WHO Health and Work Performance Questionnaire | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in objective cognitive functioning as measured by NIH Toolbox | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in disability as measured by Sheehan Disability Scale | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in subjective cognitive functioning as measured by Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Performance | From pre to post intervention (4 weeks following last intervention session, on average at 18 weeks after baseline assessment)
Change in drug cue reactivity BOLD signal in fMRI | From pre to post intervention (6 weeks following last intervention session, on average at 20 weeks after baseline assessment)
  Drug Cue Reactivity BOLD Signal is measured as average blood oxygen level dependent (BOLD) signal difference with voxel-wise analysis in the regions of interests (ROIs) (prefrontal cortex segments, cingulate cortex, insula segments, striatum nuclei, thalamus nuclei and extended amygdala nuclei) in craving > neutral contrast in drug cue exposure fMRI task with blocks of neutral and drug related images
Change in cortical-subcortical task-based connectivity in cue exposure fMRI | From pre to post intervention (6 weeks following last intervention session, on average at 20 weeks after baseline assessment)
  Cortical-subcortical task-based connectivity in cue exposure fMRI is measured as psychophysiological interaction (PPI) between average blood oxygen level dependent (BOLD) signal time series in subcortical ROIs (seeds) and voxels within prefrontal cortex and insula, using craving > neutral contrast regressor
Change in cortical-subcortical connectivity in resting state fMRI | From pre to post intervention (6 weeks following last intervention session, on average at 20 weeks after baseline assessment)
  Cortical-Subcortical Connectivity is measured as correlation between resting-state average blood oxygen level dependent (BOLD) signal time series in subcortical ROIs (seeds) and voxels within prefrontal cortex and Insula
Change in response inhibition BOLD signal in fMRI using stop signal task (SST) | From pre to post intervention (6 weeks following last intervention session, on average at 20 weeks after baseline assessment)
Change in reward processing BOLD signal fMRI using monetary incentive delay (MID) task | From pre to post intervention (6 weeks following last intervention session, on average at 20 weeks after baseline assessment)
Change in neuropsychological functioning using NIH Toolbox: Cognition | From pre to post intervention (6 weeks following last intervention session, on average at 20 weeks after baseline assessment)
  NIH toolbox: cognition includes 9 different tests: Picture Sequence Memory Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Oral Reading Recognition Test, Dimensional Change Card Sort Test, Pattern Comparison Processing Speed Test, Auditory Verbal Learning Test (Rey), Oral Symbol Digit Test. We will make a composite score using the first principal component analysis (PCA) to have one single representation of neuropsychological functioning
Drug consumption as measured with urine drug test | during intervention, 3 months, 6 months and 12 months after the intervention
  Urine drug tests for illicit drugs collected in a weekly basis summed up together during intervention, 3 months, 6 months and 12 months after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

REFERENCES:
- [Derived] Ekhtiari H, Rezapour T, Sawyer B, Yeh HW, Kuplicki R, Tarrasch M, Paulus MP, Aupperle R. Neurocognitive Empowerment for Addiction Treatment (NEAT): study protocol for a randomized controlled trial. Trials. 2021 May 7;22(1):330. doi: 10.1186/s13063-021-05268-8. PMID 33962675